CLINICAL TRIAL: NCT02042209
Title: Medical Telephone Triage of Emergency Calls for Thoracic Pain: Construction of a Probability Score for Acute Coronary Syndrome.
Brief Title: Medical Telephone Triage of Emergency Calls for Thoracic Pain
Acronym: DOREMI2
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: 0903508; PHRC interégional 2009
Record Dates: First submitted 2014-01-17; First posted 2014-01-22 (Estimated); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Acute Coronary Syndrome
Keywords: acute coronary syndrome; thoracic pain; prehospital; diagnostic score
MeSH Terms: conditions — Acute Coronary Syndrome; Chest Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Thoracic pain is the main symptom of acute coronary syndrome (ACS), urgent and serious illness. Whereas hospital mortality decreased until reaching 10%, out-of-hospital mortality remains high: half of the deaths occur during the first two hours. The benefit of an early diagnosis of ACS in term of morbidity and mortality is well established. Identification of the coronary origin of a thoracic pain by the telephone triage physician of the pre-hospital emergency service (SAMU) leads to the sending of a physician staffed ambulance (UMH) and is thus a key element of the prognosis.

The aim of the study is to build a telephone predictive score of ACS at the triage of calls for non traumatic thoracic pain. The separate analysis of the questionnaires by sex will authorize the validation of a unique score or two distinct scores for men and women.

DETAILED DESCRIPTION:
In France, approximately 30% of the calls for thoracic pain associated with an ACS do not benefit from the sending of an UMH. Our assumption is that this situation could be improved if telephone triage physicians were guided by recommendations or consensual algorithms of decision. The telephone triage doctor will manage a single questionnaire with the patient, with demographic and simple clinical data. The construction of the score will be done by the analysis of these data confronted with the final diagnosis (effective ACS or not). The effective existence of an ACS among patients with thoracic pain will be affirmed by an expert committee after collection of the intra-hospital patient's data and the follow-up at one month.

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting a non-traumatic chest pain.
* Call to the telephone triage center in first (direct call from the patient) or second intention (call of another person before the patient)

Exclusion Criteria:

- Inability to speak directly to the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years, with a non-traumatic chest pain.
Sampling Method: Non-Probability Sample
Enrollment: 4205 (Actual)
Dates: Start 2010-05; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
diagnosis of acute coronary syndrome (ACS) | one month
  The criterion selected to build these scores will be the effective existence of an ACS among included patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis DUCASSE, PH, MD, Principal Investigator — Toulouse Hospital
Locations (3):
- France (3):
  - Bordeaux Hospital Center, Bordeaux
  - La Réunion Hospital center, Saint-Denis
  - Toulouse Hosital Center, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Reuter PG, Pradeau C, Huo Yung Kai S, Lhermusier T, Bourde A, Tentillier E, Combes X, Bongard V, Ducasse JL, Charpentier S. Predicting acute coronary syndrome in males and females with chest pain who call an emergency medical communication centre. Scand J Trauma Resusc Emerg Med. 2019 Oct 17;27(1):92. doi: 10.1186/s13049-019-0670-y. PMID 31623657